CLINICAL TRIAL: NCT05737368
Title: Treatment of Recurrent Glioblastoma With Fractionated Radiotherapy Combined With Cadonilimab
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0995
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients will receive the treatment of fractionated radiotherapy and Cadonilimab (Experimental): fractionated radiotherapy (500cGy *5F, 600cGy*5F, 350cGy*10F, according to the tumor volume); within 14 days after receiving radiotherapy, Cardunizumab (10mg/kg, Q3W, d1)
  Interventions: Radiation: fractionated radiotherapy; Drug: cadonilimab

INTERVENTIONS:
Radiation: fractionated radiotherapy — fractionated radiotherapy (500cGy *5F, 600cGy*5F, 350cGy*10F, according to the tumor volume)
Drug: cadonilimab — Cardunizumab (10mg/kg, Q3W, d1)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness in the treatment of recurrent glioblastoma with Cadonilimab combined with fractionated radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. . Written and signed informed consent.
2. . Male or female, age≥ 18 and ≤ 75 years old on day of signing informed consent.
3. Epitentorial glioblastoma confirmed by pathology; Diagnosis of recurrence through clinical imaging evidence.
4. The maximum diameter of recurrent tumor is less than 6 cm.
5. Concurrent radiotherapy and chemotherapy with standard STUP treatment scheme in the past.
6. The interval from the last radiotherapy is more than 6 months.
7. KPS (Karnofsky function status score)>60.

Exclusion Criteria:

1. Prior use of investigational products or devices within 4 weeks prior to the first administration of the study treatment.
2. Concurrent enrollment into another clinical study, except the study belongs to investigational, non-interventional studies or the follow-up period of interventional studies.
3. Multiple malignant gliomas.
4. Subtentorial glioblastoma or Extracranial metastatic lesions.
5. Active autoimmune diseases.
6. Known history of primary immunodeficiency virus infection or known history of testing positive for human immunodeficiency virus (HIV).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | 3 months after treatment

SECONDARY OUTCOMES:
Local control rate (LC) | from date of enrollment to date of first documented local progression. Assessed up to 6 months
  The proportion of patients without tumor progression on imaging of brain glioma lesions was evaluated by RANO standard.
Objective Response Rate (ORR) | from date of enrollment to the date of first documented complete response or partial response. Assessed up to 6 months
  The ORR is defined as the percentage of participants having complete response or partial response to protocol treatment. Objective response will be measured by RECIST 1.1.
Disease control rate (DCR) | from date of enrollment to the date of progress. Assessed up to 6 months
  The DCR is defined as the proportion of subjects with complete response, partial response, or stable disease based on RECIST Version 1.1.
progression-free survival (PFS) | from date of enrollment to the date of first documented progression. Assessed up to 6 months
  the probability of 6-month disease progression-free survival was evaluated by RANO standard after treatment.
survival (OS) rate | from date of enrollment to the date of death from any cause. Assessed up to 6months
  Probability of survival for 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qichun Wei, MD/PhD, Study Director — Zhejiang University